CLINICAL TRIAL: NCT01914692
Title: Application of Somatostatin for Advanced Gastric Cancer After D2 Lymph Node Dissection -a Prospective Randomized Controlled Study
Brief Title: Application of Somatostatin for Advanced Gastric Cancer After D2 Lymph Node Dissection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wang Shaochuan, Postgraduate, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: nova-0426
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Gastric Cancer After D2 Lymph Node Dissection
MeSH Terms: interventions — Somatostatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Somatostatin group (Experimental): Patients with Advanced Gastric Cancer After D2 Lymph Node Dissection accept the Somatostatin medical therapy.
  Interventions: Drug: Somatostatin
- Blank group (Placebo Comparator): Use the normal saline instead of somatostatin.

INTERVENTIONS:
Drug: Somatostatin — Somatostatin is a kind of traditional medicines ,which is for the treatment of intestinal fistula，upper gastrointestinal hemorrhage.
  Arms: Somatostatin group

SUMMARY:
Gastric cancer radical surgery related complications are common.Somatostatin is a conventional medical therapy for bleeding.This study explore the effect of Somatostatin for Advanced Gastric Cancer After D2 Lymph Node dissection.

ELIGIBILITY:
Inclusion Criteria:

1. More than eighteen years old
2. Gastric cancer diagnosed by pathological examination
3. Be given informed consent
4. Without diabetes/hyperthyroidism/Damages of functions of heart, liver and kidney/Systemic Infection/immunodeficiency

Exclusion Criteria:

1. Contraindication of vascular puncture operation
2. Patients who refused to take part in the programe
3. Poor compliance of treatment
4. Malnutrition,BMI<18
5. with pancreatectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
fistula of pancreas | one year
  number of patients

SECONDARY OUTCOMES:
amount of bleeding | six months
  amount of bleeding after the operation
seroperitoneum | six months
  seroperitoneum volum of patients
infection of incisional wound | one year
  number of patients

OTHER OUTCOMES:
postoperative pancreatitis | one year
  number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Song Wu, Doctor, Study Chair — First Affiliated Hospital of Sun Yat-sen University